CLINICAL TRIAL: NCT00066482
Title: Pilot Study of Cisplatin, Etoposide, Bleomycin and Escalating Dose Cyclophosphamide Therapy for Children With High Risk Malignant Germ Cell Tumors
Brief Title: Combination Chemotherapy in Treating Children With Newly Diagnosed Malignant Germ Cell Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGCT01P1; CDR0000316244 (Other: Clinical Trials.gov)
Record Dates: First submitted 2003-08-06; First posted 2003-08-07 (Estimated); Last update posted 2013-10-17 (Estimated); Status verified 2013-10

CONDITIONS: Childhood Germ Cell Tumor; Extragonadal Germ Cell Tumor
Keywords: childhood teratoma; childhood extragonadal germ cell tumor
MeSH Terms: conditions — Teratoma | interventions — Bleomycin; Filgrastim; Granulocyte Colony-Stimulating Factor; Cisplatin; Cyclophosphamide; Etoposide; etoposide phosphate; Mesna

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- combination chemotherapy (Experimental): Induction therapy: bleomycin sulfate IV over 10-20 minutes on day 1, etoposide IV over 1 hour and cisplatin IV over 4 hours on days 1-5, and cyclophosphamide IV over 1 hour on day 1. MESNA & Filgrastim (G-CSF) subcutaneously once daily beginning on day 6 and continuing until blood counts recover. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity. 6 patients receive escalating doses of cyclophosphamide until the maximum tolerated dose (MTD) is determined.
  Evaluated after 4 courses of therapy. Partial response or stable disease undergo second-look conventional surgery & receive 2 more courses of induction therapy then re-evaluated. Those who do not achieve complete response (CR) after a total of 6 courses may undergo a third conventional surgery. Tumor that cannot be removed are removed from study therapy. Achievement of a CR at anytime are followed monthly for 1 year, every 6 months for 1 year, and then annually for 3 years.
  Interventions: Biological: bleomycin sulfate; Biological: filgrastim; Drug: cisplatin; Drug: cyclophosphamide; Drug: etoposide; Procedure: conventional surgery; Biological: MESNA

INTERVENTIONS:
Biological: bleomycin sulfate — Given IV over 10 minutes. Children ≥ 12 months: 15 units/m2/dose Children < 12 months: 0.5 units/kg/dose Day 1 (Week 1, 4, 7, 10)
  Other Names: BLEO; BLM; Blenoxane; NSC #125066
Biological: filgrastim — Given SQ once daily 5 micrograms/kg/dose Starting on Day 6 (Week 1, 4, 7, 10) Daily until ANC > 5,000/uL
  Other Names: GRANULOCYTE COLONY-STIMULATING FACTOR; r-metHuG-CSF; G-CSF; Neupogen; NSC #614629
Drug: cisplatin — Children ≥ 12 months: Given IV over one hour Dose: 20 mg/m2/dose Days 1-5 (Week 1,4,7,10) Children < 12 months: Given IV over 4 hours, 0.67 mg/kg/dose Days 1-5 (Week 1,4,7,10)
  Other Names: Cis-diamminedichloroplatinum II; Platinol-AQ; NSC #119875
Drug: cyclophosphamide — Given IV over 1 hour. Children ≥ 12 months: Level 1: 1.2 g/m2/dose Level 2: 1.8 g/m2/dose Level 3: 2.4 g/m2/dose Children < 12 months: Level 1: 40 mg/kg/dose Level 2: 60 mg/kg/dose Level 3: 80 mg/kg/dose Day 1 (Week 1, 4, 7, 10)
  Other Names: Cytoxan; NSC #026271
Drug: etoposide — Given IV over 1 hour. Children ≥ 12 months: 100 mg/m2/dose Children < 12 months: 3.3 mg/kg/dose Day 1-5 (Week 1, 4, 7, 10)
  Other Names: VP-16; VePesid; Etopophos; NSC #141540
Procedure: conventional surgery — Stage III/IV extragonadal tumors: biopsy followed by a definitive surgical excision after maximal chemotherapy effect, likely after 4 cycles of therapy
Biological: MESNA — Given IV or oral. The total daily MESNA dose is equal to at least 80% of the daily CPM dose. The oral dose of MESNA is 2x the IV dose. Day 1 (Week 1,4,7,10) To be given with CPM.
  Other Names: sodium 2-mercaptoethane sulfonate; Mesnex; NSC #113891

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effect on the body of combining cyclophosphamide with cisplatin, etoposide, and bleomycin in treating children who have newly diagnosed malignant germ cell tumors that are not in the brain and gonads.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose and toxicity profile of cyclophosphamide in combination with bleomycin, etoposide, and cisplatin in pediatric patients with newly diagnosed high-risk extracranial, extragonadal malignant germ cell tumors.
* Determine the response rate in patients treated with this regimen.

OUTLINE: This is a pilot, multicenter, dose-escalation study of cyclophosphamide.

* Induction therapy: Patients receive bleomycin IV over 10-20 minutes on day 1, etoposide IV over 1 hour and cisplatin IV over 4 hours on days 1-5, and cyclophosphamide IV over 1 hour on day 1. Patients also receive filgrastim (G-CSF) subcutaneously once daily beginning on day 6 and continuing until blood counts recover. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 6 patients receive escalating doses of cyclophosphamide until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

Patients are evaluated after 4 courses of therapy. Patients with partial response or stable disease undergo second-look surgery, receive 2 more courses of induction therapy, and are then re-evaluated. Patients who do not achieve complete response (CR) after a total of 6 courses may undergo a third surgery. Patients who still have tumor that cannot be removed are removed from study therapy. Patients who achieve a CR at anytime are followed.

Patients are followed monthly for 1 year, every 6 months for 1 year, and then annually for 3 years.

PROJECTED ACCRUAL: A total of 6-18 patients will be accrued for this study within 1.3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed newly diagnosed extracranial germ cell tumors, including 1 of the following types:

  * Yolk sac carcinoma (endodermal sinus tumor)
  * Embryonal carcinoma
  * Choriocarcinoma
  * Teratoma with mixed malignant elements (malignant teratoma)
* High-risk disease, defined as stage III or IV extragonadal germ cell tumors
* Must be enrolled on study within 21 days of diagnostic surgical procedure

PATIENT CHARACTERISTICS:

Age

* 21 and under (at original diagnosis)

Performance status

* ECOG 0-2

  * Karnofsky 50-100% (in patients over 16 years of age)
  * Lansky 50-100% (in patients 16 years of age and under)

Life expectancy

* At least 2 months

Hematopoietic

* Absolute neutrophil count at least 1,000/mm^3
* Platelet count at least 100,000/mm^3 (transfusion independent)
* Hemoglobin at least 10.0 g/dL (transfusion allowed)

Hepatic

* Not specified

Renal

* Creatinine clearance or radioisotope glomerular filtration rate at least 70 mL/min OR
* Creatinine based on age as follows:

  * No greater than 0.8 mg/dL (5 years and under)
  * No greater than 1.0 mg/dL (6-10 years)
  * No greater than 1.2 mg/dL (11-15 years)
  * No greater than 1.5 mg/dL (over 15 years)

Pulmonary

* FEV_1/FVC greater than 60% OR
* Children who are uncooperative must meet all of the following criteria:

  * No dyspnea at rest
  * No exercise intolerance
  * Pulse oximetry greater than 94%

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy

Surgery

* See Disease Characteristics

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2004-07; Primary Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Feasibility of adding cyclophosphamide to a PEB backbone | 2 years

SECONDARY OUTCOMES:
Maximum tolerated dose | 21 days
  Maximum tolerated dose (MTD) and toxicity profile of cyclophosphamide combined with cisplatin, etoposide, bleomycin (C-PEB) in previously untreated children with high-risk malignant germ cell tumors (MGCT).
Estimate the response rate | Length of study
  To estimate the response rate in this group of patients to a regimen of cyclophosphamide combined with cisplatin, etoposide, bleomycin (C-PEB).

CONTACTS AND LOCATIONS:
Overall Officials: Marcio A. Malogolowkin, MD, Study Chair — Children's Hospital Los Angeles
Locations (98):
- United States (88):
  - Comprehensive Cancer Center at University of Alabama at Birmingham, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Southern California Permanente Medical Group, Downey, California
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - Children's Hospital of Orange County, Orange, California
  - Kaiser Permanente Medical Center - Oakland, Sacramento, California
  - Children's Hospital and Health Center - San Diego, San Diego, California
  - Stanford Cancer Center at Stanford University Medical Center, Stanford, California
  - Children's Hospital Cancer Center, Denver, Colorado
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lee Cancer Care of Lee Memorial Health System, Fort Myers, Florida
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Miami Children's Hospital, Miami, Florida
  - Baptist-South Miami Regional Cancer Program, Miami, Florida
  - Sacred Heart Cancer Center at Sacred Heart Hospital, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - St. Joseph's Cancer Institute at St. Joseph's Hospital, Tampa, Florida
  - Kaplan Cancer Center at St. Mary's Medical Center, West Palm Beach, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - St. Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - CancerCare of Maine at Eastern Maine Medial Center, Bangor, Maine
  - Alvin and Lois Lapidus Cancer Institute at Sinai Hospital, Baltimore, Maryland
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - C.S. Mott Children's Hospital at University of Michigan, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Spectrum Health Cancer Care - Butterworth Campus, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Breslin Cancer Center at Ingham Regional Medical Center, Lansing, Michigan
  - Children's Hospital of Minnesota - Minneapolis, Minneapolis, Minnesota
  - Fairview University Medical Center - University Campus, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Children's Mercy Hospital, Kansas City, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - Hackensack University Medical Center Cancer Center, Hackensack, New Jersey
  - St. Barnabas Medical Center, Livingston, New Jersey
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Medical Center - Dayton, Dayton, Ohio
  - Tod Children's Hospital - Forum Health, Youngstown, Ohio
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Greenville Hospital System Cancer Center, Greenville, South Carolina
  - East Tennessee Children's Hospital, Knoxville, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Texas Tech University Health Sciences Center School of Medicine, Amarillo, Texas
  - Children's Hospital of Austin, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - Baylor University Medical Center - Houston, Houston, Texas
  - M.D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - INOVA Fairfax Hospital, Fairfax, Virginia
  - Carilion Cancer Center of Western Virginia, Roanoke, Virginia
  - West Virginia University - Robert C. Byrd Health Sciences Center - Charleston Division, Charleston, West Virginia
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Princess Margaret Hospital for Children, Perth, Western Australia, Australia
- Canada (8):
  - Children's & Women's Hospital of British Columbia, Vancouver, British Columbia
  - Janeway Children's Health and Rehabilitation Centre, St. John's, Newfoundland and Labrador
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Montreal Children's Hospital at McGill University Health Center, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Ste-Foy, Quebec
  - Allan Blair Cancer Centre at Pasqua Hospital, Regina, Saskatchewan
- San Jorge Children's Hospital, Santurce, Puerto Rico